CLINICAL TRIAL: NCT05554445
Title: Observational Investigation of the CDED in a Real World IBD Clinic: Dietician and Patient Adaptations to the Dietary Protocol
Brief Title: Observational Investigation of the CDED in a Real World IBD Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eli Sprecher, MD (Other Government)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, Head of R&D, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: 0225-21-TLV
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult CD patients who are prescribed the Crohn disease exclusion diet: Clinically stable CD patients with active disease by CD symptoms score 4 <Harvey-Bradshaw index (HBI) at baseline and Calprotectin>50g/l / endoscopy / imaging proven active disease from the previous 4 months

SUMMARY:
A prospective observational study, which will follow a cohort of adult CD patients who are prescribed the Crohn disease exclusion diet (CDED) during their routine clinical dietary therapy. The diet is composed of three phases, at the end of the first two phases we will evaluate whether the patient achieved remission and at the end of phase three the maintenance of remission. We intend to study achievement and remission rate in association to the diet adaptations made by dieticians at phase 1 and 2, together with patient's choice off food at the third phase under real world clinical setting and patient lifestyle characteristics.

DETAILED DESCRIPTION:
This is a prospective observational study that will follow a cohort of CD patients who are prescribed the Crohn disease exclusion diet (CDED) during their routine clinical dietary therapy at the IBD clinic of the TLVMC. The CD exclusion diet (CDED), is a whole-food diet designed to reduce exposure to dietary components, hypothesized to negatively affect the microbiome (dysbiosis), intestinal barrier, and intestinal immunity. We intend to follow patients with proven clinically active disease from the previous 4 months. Disease activity will be determined by Harvey-Bradshaw index (4<HBI<16) and Calprotectin>50g.

The diet is composed of three phases, the first two included 5 mandatory foods consumed daily to provide specific fibers and starches as substrates for short chain fatty acids-producing taxa from Firmicutes, as well as sources of lean protein that were low in animal fat to decrease Proteobacteria and improve intestinal permeability, while maintaining a balanced diet. The diet included avoidance or reduction of exposure to foods containing animal/dairy fat, high fat from other sources, wheat, red or processed meat and protein sources rich in taurine, emulsifiers, artificial sweeteners, carrageenans and sulfites. The second phase stepdown diet involves higher exposure to fruits, vegetables, and legumes along with some foods that are reintroduced with restrictions to increase food flexibility and relieve monotony. The third phase of the study, is considered a maintenance phase in which patients are advised to continue practicing the concepts of the previous two phases, but they may generally manage their diet freely.

In this observational study, we aim to describe our real-world experience with the CDED, in a tertiary referral center for IBD patients. We aim to characterize both the adaptations of the first two phases of the diet practiced by IBD dieticians, and the food choices made by patients during the third phase of the diet . We aim to associate both these determinants with clinical remission at the end of phase two and remission maintenance at the end of phase three respectively.

Data collection

Upon visits, patients will be asked to fill in food frequency questionnaire (FFQ), 3-days recall questionnaires, food related quality of life, CD symptom and pain questionnaire. Dieticians will be asked to meticulously describe the adaptations they have performed in the CDED and the reasons for them at baseline, week 6 and 12. The adaptation will be made in accordance to patient's symptoms and disease characteristics.

At each visit, patient will provide a fecal sample which will be used to test for calprotectin, a biochemical marker, specific for intestine inflammation. Together with Harvey-Bradshaw index (HBI) we will determine disease severity and activity levels. Fecal sample will also use to determine and monitor changes in microbiome composition.

Anthropometric and nutritional evaluation

Patient's weight (kg), height (m), waist circumference (cm) will be documented at each study visit, and body mass index (BMI) will be calculated. Handgrip strength will be measured by a handgrip dynamometer (JAMAR® hydraulic hand dynamometer), and body composition by body electrical impedance (INBODY diagnostic weight).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Clinically stable CD patients, constant medicinal regimen throughout the study period. Refractory to mesalamine at least 6 weeks, or steroids at least 2 week, or immunomodulator at least 12 weeks or biologics at least 12 weeks therapy, medical cannabis at least 2 weeks before the study.
3. Clinically active disease by CD symptoms score 4 <Harvey-Bradshaw index (HBI) at baseline and Calprotectin>50g/l / endoscopy / imaging proven active disease from the previous 4 months.

Exclusion Criteria:

1. Inability to sign informed consent and complete study protocol
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CD patients who are prescribed the CDED during their routine clinical dietary therapy at the IBD clinic of the TLVMC.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rates will be measured by Harvey-Bradshaw Index at the end of phase 1 | week 6, end of phase 1
  Achievement of clinical remission by the end of the first phase of the diet, will be defined as HBI(Harvey-Bradshaw Index)<4
Clinical remission rates will be measured by Harvey-Bradshaw Index at the end of phase 2 | week 12, end of phase 2
  Achievement of clinical remission by the end of the second phase of the diet will be defined as HBI(Harvey-Bradshaw Index)<4
Rate of patients maintaining clinical remission at the end of phase 3 | week 24, end of phase 3
  Maintaining clinical remission by the end of the third phase of the diet will be defined as HBI(Harvey-Bradshaw Index)<4

SECONDARY OUTCOMES:
Associations between adaptations of the first phase of the diet practiced by IBD dieticians and clinical remission | week 6
  We aim to characterize the adaptations of the first phase of the diet practiced by IBD dieticians and associate the adaptations with achieving clinical remission at the end of phase 1.
  Dieticians will be asked to meticulously describe the adaptations they have performed in the CDED and the reasons for them at baseline (table 1). A 3 day food diary will be analyzed and associate with achieving remission.
  Remission will be determined by HBI<4
Associations between adaptations of the second phase of the diet practiced by IBD dieticians and clinical remission | week 12
  Dieticians will be asked to meticulously describe the adaptations they have performed to the second phase of the diet and the reason for them.
  Food diary will be analyzed and associate with achieving remission by the end of phase 2.
  Remission will be determined by HBI (Harvey-Bradshaw Index)<4
Associations between food choices during the third phase of the diet made by patients and remission maintenance | week 24
  We aim to characterize the food choices during the third phase of the diet made by patients and its association with maintaining remission at the end of phase 3.
  Food choice will be analyzed according to Food frequency questionnaire (FFQ) and food dairy and associate with maintaining remission.
  Remission will be determined by HBI (Harvey-Bradshaw Index)<4

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Tel Aviv Medical Center- Head of Inflammatory Bowel Disease Center
Locations (2):
- Israel (2):
  - Department of Gastroentherology,Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Sourasky medical center (Ichilov), Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
As part of future collaboration between researchers, all medical information and fecal samples would be transferred in an anonymous manner (it will not include any identifying detalis to partners outside the hospital), and in accordance with a contract approved by the hospital's research and development department.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After termination of the study protocol for all participants
Access Criteria: Medical information and fecal samples would be transferred in an anonymous manner, with no identifying details of the patients